CLINICAL TRIAL: NCT05420558
Title: The Application of Molecular Probe Targeting Fibroblast Activation Protein in Malignant Tumor of Digestive System
Brief Title: Fibroblast Activation Protein Inhibitor PET/CT Imaging in Malignant Tumor of Digestive System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZNYYPTXM2022013
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Gastrointestinal Cancer
Keywords: fibroblast activation protein inhibitor; positron emission tomography; gastrointestinal cancer; digestive system tumor; recurrence; metastases; prognosis
MeSH Terms: conditions — Gastrointestinal Neoplasms; Digestive System Neoplasms; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fibroblast activation protein inhibitor PET/CT imaging — All participants will receive a 68Ga-labelled fibroblast activation protein inhibitor PET/CT imaging

SUMMARY:
The purpose of this single center prospective study is to assess the value of FAPI PET imaging in predicting early postoperative recurrence of malignant tumor of digestive system and to evaluate the diagnostic performance of FAPI PET/CT in the detection of primary tumor and metastatic lesions.

DETAILED DESCRIPTION:
Malignant tumor of digestive system is one of the most common cancer types worldwide with high cancer-related mortalities. FDG PET/CT is an essential imaging modality in the tumor treatment and management. However, FDG PET/CT has certain limitations. For example, the detection sensitivity and tracer uptake in signet ring cell carcinoma (SRCC) is low. Furthermore, the physiological uptake of the gastrointestinal tract and acute gastroenteritis may mask the detection of lesion in the abdomen and pelvis. Therefore, a novel molecular imaging tracer is needed for the accurate evaluation of malignant tumor of digestive system.

Cancer-associated fibroblasts (CAFs) specifically express fibroblast activation protein (FAP), which is highly expressed by CAFs in more than 90% of human epithelial cancers. FAP-specific small molecule inhibitors (FAPIs) show much advantages over FDG, including high tumor accumulation, low background tissue uptake, and rapid clearance in vivo.

The purpose of this single center prospective study is to assess the value of FAPI PET/CT imaging in predicting early postoperative recurrence of malignant tumor of digestive system and to evaluate the diagnostic performance of FAPI PET/CT in the detection of primary tumor and metastatic lesions.

In this study, qualitative and quantitative analyses will be used. The diagnostic criteria of FAPI PET/CT: if the FAPI uptake of lesion is higher than that of the surrounding background tissue, it is determined as a positive lesion; if the FAPI uptake of the lesion is the same as or lower than that of the surrounding background tissue, it is determined as a negative lesion. Pathological result is used as the gold standard for diagnosis. The diagnostic performance of FAPI PET/CT including sensitivity, specificity, positive predictive value, negative predictive value, and accuracy will be calculated.

The quantitative indicators include the following metabolic parameters: maximum standard uptake value (SUVmax), mean standard uptake value (SUVmean), tumor metabolic volume (MTV), total tumor glycolysis (TLG), tumor-to-liver ratio, and tumor-to-background tissue ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign the informed consent.
2. Patients with suspected or new diagnosed gastrointestinal cancer or other malignant tumor of digestive system.
3. Complete clinical information, biochemical examination results, CT and/or MRI imaging examination, pathological information, and clinical/imaging follow-up data.

Exclusion Criteria:

1. Female patient who plan to become pregnant within 6 months, or pregnant or breast-feeding women.
2. Allergic constitution.
3. Those who are in poor general condition and cannot tolerate PET/CT examination.
4. The researchers believe that he or she is not suitable to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or new diagnosed gastrointestinal cancer or other malignant tumor of digestive system.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
early postoperative recurrence | two years
  Evaluation of the value of FAPI PET imaging in predicting early postoperative recurrence of malignant tumor of digestive system

SECONDARY OUTCOMES:
diagnostic performance | 18 months
  Evaluation of the diagnostic performance of FAPI PET imaging in detecting malignant tumor of digestive system

CONTACTS AND LOCATIONS:
Overall Officials: Chongjiao Li, MD, PhD, Study Director — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared with other researchers. Our research results will eventually be shared with other researchers in the form of paper.

REFERENCES:
- [Background] Lin R, Lin Z, Chen Z, Zheng S, Zhang J, Zang J, Miao W. [68Ga]Ga-DOTA-FAPI-04 PET/CT in the evaluation of gastric cancer: comparison with [18F]FDG PET/CT. Eur J Nucl Med Mol Imaging. 2022 Jul;49(8):2960-2971. doi: 10.1007/s00259-022-05799-5. Epub 2022 Apr 25. PMID 35462566
- [Background] Fu L, Huang S, Wu H, Dong Y, Xie F, Wu R, Zhou K, Tang G, Zhou W. Superiority of [68Ga]Ga-FAPI-04/[18F]FAPI-42 PET/CT to [18F]FDG PET/CT in delineating the primary tumor and peritoneal metastasis in initial gastric cancer. Eur Radiol. 2022 Sep;32(9):6281-6290. doi: 10.1007/s00330-022-08743-1. Epub 2022 Apr 5. PMID 35380229
- [Background] Qin C, Song Y, Gai Y, Ruan W, Liu Q, Liu F, Zheng D, Zhang P, Liu H, Zhang T, Tao K, Lan X. Gallium-68-labeled fibroblast activation protein inhibitor PET in gastrointestinal cancer: insights into diagnosis and management. Eur J Nucl Med Mol Imaging. 2022 Oct;49(12):4228-4240. doi: 10.1007/s00259-022-05847-0. Epub 2022 Jun 3. PMID 35657428